CLINICAL TRIAL: NCT02582411
Title: Laser Speckle Flowgraphy in Caucasians: Age Dependence and Comparison With Doppler Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Other Study IDs: OPHT-040415
Record Dates: First submitted 2015-10-07; First posted 2015-10-21 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Group 1: 18-34 years: Patients in age group 18-34 years
  Interventions: Device: Laser Speckle Flowgraphy; Device: Doppler Optical Coherence Tomography
- Group 2: 35-49 years: Patients in age group 35-49 years
  Interventions: Device: Laser Speckle Flowgraphy
- Group 3: 50-64 years: Patients in age group 50-64 years
  Interventions: Device: Laser Speckle Flowgraphy
- Group 4: 65-80 years: Patients in age group 65-80 years
  Interventions: Device: Laser Speckle Flowgraphy

INTERVENTIONS:
Device: Laser Speckle Flowgraphy — A commercially available LSFG (Softcare, Fukutsu, Japan) system will be used in the present study. The LSFG device consists of a fundus camera equipped with a diode laser with a wavelength if 830 nm and charge-coupled device. NB, the relative velocity of blood flow, is derived from the pattern of speckle contrast produced by the interference of a laser scattered by blood cells moving in the ocular fundus. Images are acquired continuously at the rate of 30 frames per seconds in a 4-second time period and stored on a personal computer. Heartbeat map of the optic nerve head and the retina/choroid is generated
  Other Names: LSFG
Device: Doppler Optical Coherence Tomography — A dual-beam bidirectional Doppler OCT system comprises a broadband superluminescent diode (SLD) with a central wavelength of 840 (spectral bandwidth 54 nm) and two CCD cameras with a maximum readout rate of 20 kHz. The system provides a resolution (in tissue) of about 6 and 18 μm in axial and lateral direction, respectively. The sample, i.e. the retinal vessel under study, is illuminated by two probe beams separated by their polarization properties. Light back scattered and backreflected from the sample is spectrally detected by two identical spectrometers and postprocessing, i.e.
  calculation the phase shift due moving scatterers within the sample, is carried out by a personal computer with software written in National Instruments LabView. The power of both probe beams incident on the cornea is 650 μW, which is below the ANSI (American National Standard Institute) limits for small source ocular exposure to a laser beam within the measuring time.
  Groups: Group 1: 18-34 years

SUMMARY:
Some of the most prevalent eye diseases such as age-related macular degeneration, glaucoma and diabetic retinopathy are associated with ocular perfusion abnormalities. Currently, there is no gold-standard method for the measurement of ocular blood flow available. Laser speckle flowgraphy is a promising technique for the two-dimensional assessment of ocular blood flow in humans. So far the technique has, however, been only gained widespread use in Japan. The experience in Caucasian subjects is very limited. In a Japanese population it was shown that mean blur rate, a measure of chorioretinal blood velocity, decreases with age. This is of relevance, because an age-related decline in ocular blood flow may partially explain the age-dependence of ocular vascular disease. The present study investigates this age-dependence in healthy subjects. In addition, the investigators investigate in a sub-group of this population whether relative flow volume (RFV), a novel index of blood flow in the human retina derived from laser speckle flowgraphy is associated with retinal blood flow as assessed with bi-directional Doppler Optical Coherence Tomography (DOCT).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years, nonsmokers
* Subject is generally healthy with no current significant or a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination. A significant disorder is defined as a disease or medical condition associated with impaired health status, requiring regular or current medical treatment and/or follow up. For the purposes of this study, an investigator may classify a medical condition as a nonsignificant disorder despite the fact that the subject receives treatment. Subjects having controlled Stage 1 hypertension (blood pressure of 140-159 mmHg systolic and/or 90- 99 mmHg diastolic) are eligible for participation in this study.
* Normal ophthalmic findings, ametropia < 6 Dpt

Exclusion Criteria:

* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Wearing of contact lenses
* Ocular infection or clinically significant inflammation
* Ocular surgery in the 3 months preceding the study
* Blood donation in the 3 weeks preceding the study
* Pregnancy, planned pregnancy or lactating
* Opacities of the cornea (e.g. corneal scars, corneal oedema), the lens (e.g. Lens opacities classification system version II (LOCS-II) grading > 2, posterior capsule opacification) or the vitreous (e.g. vitreous haemorrhage, asteroid hyalosis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 healthy subjects in 4 age groups Group 1: 18-34 years Group 2: 35-49 years Group 3: 50-64 years Group 4: 65-80 years
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Relative flow volume (LSFG) | 3 weeks

SECONDARY OUTCOMES:
Systemic blood pressure | 3 weeks
Intraocular pressure | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Luft N, Wozniak PA, Aschinger GC, Fondi K, Bata AM, Werkmeister RM, Schmidl D, Witkowska KJ, Bolz M, Garhofer G, Schmetterer L. Measurements of Retinal Perfusion Using Laser Speckle Flowgraphy and Doppler Optical Coherence Tomography. Invest Ophthalmol Vis Sci. 2016 Oct 1;57(13):5417-5425. doi: 10.1167/iovs.16-19896. PMID 27756076